CLINICAL TRIAL: NCT03252418
Title: Ascorbic Acid Versus Diode Laser in the Treatment of Gingival Hyperpigmentation: Histological and Clinical Randomized Study
Brief Title: Ascorbic Acid Versus Diode Laser in the Treatment of Gingival Hyperpigmentation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dalia Yosri, Assistant lecturer of oral medicine and periodontology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDASU-RECIM10201512
Record Dates: First submitted 2017-08-15; First posted 2017-08-17 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Gingival Hyperpigmentaion
Keywords: ascorbic acid; diode laser; gingival hyperpigmentation
MeSH Terms: interventions — Ascorbic Acid; Lasers, Semiconductor

STUDY DESIGN:
Intervention Model Description: treating of gingival hyperpigmentation by two different methods
Who Masked: Outcomes Assessor
Masking Description: when measuring the gingival brightness and MAF of melanosomes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ascorbic acid (Experimental): injection of 1 ml intamucosal ascorbic acid 3 times with 1 week interval
  Interventions: Drug: Ascorbic Acid 500 MG
- diode laser (Experimental): photothermolysis by diode laser in one session
  Interventions: Device: diode laser

INTERVENTIONS:
Drug: Ascorbic Acid 500 MG — ascorbic acid is vitamin that can cause gingival depigmentation
  Arms: ascorbic acid
Device: diode laser — diode laser is soft tissue laser case photothermolysis of melanoctes
  Arms: diode laser

SUMMARY:
Vitamin C affect the melanocytes function not the number while diode laser cause melanocytes destruction. Although diode laser and vitamin C have proved their effectiveness in depigmentation in previous studies, there are no published studies compared the effect of diode laser and vitamin C on melanocytes and melanosomes clinically and histologically.

DETAILED DESCRIPTION:
Cosmetic dentistry is usually centered on aesthetic restorative procedures but it may also involve the appearance of the gingiva, especially when it is located in the anterior labial region. Oral pigmentation may be physiological or pathological in nature. Better esthetics results of depigmentation were achieved with diode laser than conventional scalpel and with rotary abrasion, also diode laser is effective and safe in removal of gingival hyperpigmentation and repigmentation doesn't occur.When choosing a depigmenting agent, it is important to differentiate between substances that are toxic to the melanocyte and substances that interrupt the key steps of melanogenesis. Vit. C interacts with copper ions at the tyrosinase-active site and inhibits action of the enzyme tyrosinase, thereby decreasing the melanin formation.

This randomized comparative clinical study was conducted on ten patients attending the outpatient clinic of the Oral Medicine and Periodontology department, Faculty of Dentistry, Ain Shams University and seeking treatment for their gingival hyperpigmentation for esthetic reason.

The study was conducted after receiving an ethical clearance from the Research Ethics Committee of Ain Shams University, Faculty of Dentistry; that the study follows the ethical guidelines of research. The patients clearly understood the purpose of this study and signed an informed consent.

According to the study results, vit C treated patients showed no or little repigmentation after six months post treatment. Conversely, diode laser treated patients showed significant recurrence of gingival pigmentation after six months post treatment. These could be attributed to the blocking effect of vitamin C on the existing melanocytes to form new melanoseomes, however diode laser cause removal of the existing melanocytes that may cause formation of new melanocytes (migrating from neighboring melanocytes from the adjacent area of the gingiva) with the ability of forming new melanosomes and causing repigmentation. Histopathological assessment revealed that both treatment modalities caused significant reduction in MAF after six months post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with age ranging from 18 years old to 40 years old.
* Bilaterally symmetric gingival hyperpigmentation on the maxillary and mandibular labial keratinized gingiva between canines.
* Patients free from any systemic diseases as evidenced by the health questionnaire, using modified Cornell medical index (Pendleton et al., 2004).
* Patients with thick gingival biotype ≥ 3 mm.

Exclusion Criteria:

* Presence of local condition that may cause gingival hyperpigmentation (traumatized epithelium caused by defective fixed prosthesis or restoration).
* Smokers.
* Pregnant or lactating females.
* Patients with poor oral hygiene, incompliance to treatment and persistence gingival inflammation after phase I periodontal therapy.
* Clinically diagnosed periodontitis (attachment and bone loss, presence of periodontal pockets, gingival recession and tooth mobility).
* Previous treatment to pigmentation.
* Patients taking supplementary vitamin C for any reason.
* Known sensitivity to ascorbic acid or any of its derivatives.
* Patients taking any drug that may cause gingival pigmentation.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-10-07 (Actual); Primary Completion 2016-09-10 (Actual); Study Completion 2016-09-10 (Actual)

PRIMARY OUTCOMES:
Dummett oral pigmentaion index (DOPI) | change from baseline to 1, 3 and 6 months
  scoring from 0 ( no pigmentation to 3 (sever pigmentation
gingival brightness (ΔL) | change from baseline to 1, 3 and 6 months
  using spectrophotometer
histological mean area fraction of melanosomes | change from baseline to 6 months
  by taking soft tissue samples and stained by fontana masson stain

SECONDARY OUTCOMES:
patient satisfaction questionnaire | immediate postopearive, 1 week, 1 month and 6 months
  from scoring patients pain and cosmetic changes

CONTACTS AND LOCATIONS:
Overall Officials: Nevine H kheir ElDien, Professor, Study Director — faculty of Dentistry- Ain Shams univesity